CLINICAL TRIAL: NCT04849364
Title: A Phase II Circulating Tumor DNA Enriched, Genomically Directed Post-neoadjuvant Trial for Patients With Residual Triple Negative Breast Cancer (PERSEVERE)
Brief Title: Circulating Tumor DNA Enriched, Genomically Directed Post-neoadjuvant Trial for Patients With Residual Triple Negative Breast Cancer
Acronym: PERSEVERE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funder Decision
Sponsor: Bryan Schneider, MD (Other)
Collaborators: Genentech, Inc. (Industry); Pfizer (Industry); Foundation Medicine (Industry); Indiana University (Other); Vera Bradley Foundation for Breast Cancer (Other)
Responsible Party: Sponsor-Investigator, Bryan Schneider, MD, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCRN BRE18-334
Record Dates: First submitted 2021-04-13; First posted 2021-04-19 (Actual); Results first posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Capecitabine; talazoparib; pembrolizumab; inavolisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): Arm 1a: Patients who are ctDNA-positive and harbor a genomic target. DNA repair pathway = talazoparib + capecitabine (CLOSED)
  Arm 1b: Patients who are ctDNA-positive and harbor a genomic target. Immunotherapy pathway = pembrolizumab + capecitabine (CLOSED)
  Arm 1c: Patients who are ctDNA-positive and harbor a genomic target. PI3K Pathway = inavolisib + capecitabine ---> +/- standard of care pembrolizumab
  Arm 1d: Patients who are ctDNA-positive and harbor a genomic target. DNA Repair + Immunotherapy = talazoparib + capecitabine +/- standard of care pembrolizumab
  Interventions: Drug: Capecitabine; Drug: Talazoparib; Drug: Pembrolizumab; Drug: Inavolisib
- Arm 2 (Active Comparator): Arm 2 subjects have plasma ctDNA positive but do not have a genomically driven treatment option. Treatment of physician's choice will be given with consideration for capecitabine and pembrolizumab. Dose, schedule and duration of treatment to be determined by treating physician.
  Interventions: Drug: Capecitabine; Drug: Pembrolizumab
- Arm 3 (Active Comparator): Arm 3 subjects have plasma ctDNA negative. Treatment of patient and physician's choice will be given with consideration for capecitabine and pembrolizumab. Dose, schedule and duration of treatment to be determined by treating physician.
  Interventions: Drug: Capecitabine; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Capecitabine — Capecitabine 1000 mg/m2 BID Orally 14 days on and 7 days off Cycle = 21 days; Total of 8 cycles
  Other Names: Xeloda
Drug: Talazoparib — Talazoparib Cycle 1: 0.75 mg then Cycle 2-8: 1 mg Cycle = 21 days; Total of 8 cycles
  Other Names: Talzenna
  Arms: Arm 1
Drug: Pembrolizumab — Per standard of care.
  Other Names: Keytruda
Drug: Inavolisib — Inavolisib Cycle 1: 6 mg then Cycle 2-8: 9mg Orally 21 days on Cycle = 21 days; Total of 8 cycles
  Other Names: GDC-0077
  Arms: Arm 1

SUMMARY:
This is a 3-arm study stratified by plasma ctDNA. Patients with residual TNBC disease after pre-operative therapy will be assigned to 1 of 3 Arms based on plasma ctDNA positivity and genomic marker(s).

DETAILED DESCRIPTION:
Participants that are plasma ctDNA positive with a genomic target will be assigned to one of the three groups in Arm 1 and receive genomically directed therapy.

* Arm 1a: DNA Repair pathway = talazoparib + capecitabine (CLOSED)
* Arm 1b: Immunotherapy pathway = pembrolizumab + capecitabine (CLOSED)
* Arm 1c: PI3K Pathway = inavolisib + capecitabine ---> +/- standard of care pembrolizumab
* Arm 1d: DNA Repair + Immunotherapy = talazoparib + capecitabine +/- standard of care pembrolizumab

Participants that are plasma ctDNA positive without a genomic target will be assigned to Arm 2 and receive capecitabine and pembrolizumab or treatment of physician's choice.

Participants that are plasma ctDNA negative will be assigned to Arm 3 and receive any of the following based on patient and physician decision: no therapy/observation, capecitabine and pembrolizumab or treatment of physician's choice.

ELIGIBILITY:
General Inclusion Criteria

* Written informed consent and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or may be obtained separately.
* Age ≥ 18 years at the time of consent.
* ECOG Performance Status 0 or 1 within 28 days prior to study registration.
* Must have histologically or cytologically confirmed triple negative (ER-/PR-/HER2-) invasive breast cancer per pathology report. NOTE: ER and PR will be considered negative if ≤ 10% of cells stain weakly positive. HER2 will be considered negative if scored 0 or 1+ by immunohistochemistry (IHC) or 2+ by IHC associated with a fluorescence in situ hybridization (FISH) ratio of < 2.0 or < 6 copies per cell.
* Must have clinical stage I-III at diagnosis (AJCC 8th edition) based on initial evaluation by physical examination and/or breast imaging prior to neoadjuvant chemotherapy.
* Must have completed preoperative (neoadjuvant) chemotherapy for this index case. NOTE: Acceptable preoperative regimens include an anthracycline or a taxane, or both. Participants who received preoperative therapy as part of a clinical trial may enroll. Participants may not have received adjuvant chemotherapy after surgery prior to registration. Bisphosphonate use is allowed.
* Subjects who received pembrolizumab in the neoadjuvant setting are eligible and may continue treatment during the screening process. Subjects assigned to Arm 1 will require a 3 week wash out period prior to initiation of study treatment. Subjects may resume pembrolizumab to complete the planned year of therapy (17 cycles) after completion of study therapy based on investigator discretion. Subjects assigned to Arm 2 and Arm 3 may continue pembrolizumab treatment during the study based on investigator discretion. Total duration of pembrolizumab treatment should not be extended beyond 17 cycles.
* Must have significant residual invasive disease at the time of definitive surgery following preoperative chemotherapy. Significant residual disease is defined as at least one of the following:

  * Residual invasive disease in the breast measuring at least 1 cm. The presence of DCIS without invasion does not qualify as residual disease in the breast.
  * Any macroscopic, (≥ 2mm) residual, lymph node involvement regardless of primary tumor site involvement (includes no residual disease in the breast).
  * Residual cancer burden (RCB) score 2 or 3.
* Must have completed definitive resection of primary tumor. Participants must begin assigned arm therapy no later than 96 days from the last local therapy. NOTE: Negative margins for both invasive and ductal carcinoma in situ (DCIS) are desirable, however participants with positive margins may enroll if the study site treatment team believes no further surgery is possible and participant has received radiotherapy. Participants with margins positive for lobular carcinoma in situ (LCIS) are eligible. Either mastectomy or breast conserving surgery (including lumpectomy or partial mastectomy) is acceptable.
* Breast Radiotherapy

  * Radiotherapy is required for participants who underwent breast-conserving therapy, including lumpectomy or partial mastectomy unless deemed inappropriate by the treating provider.
  * Post mastectomy radiation is at the discretion of the treating physician.
  * If radiation was given prior to surgery, additional radiation after surgery is not required.
  * In all cases participants must begin arm assigned therapy no later than 96 days from the last local therapy
  * Any acute toxicity must have resolved to grade < 2 prior to starting arm specific therapy.
* Must consent to allow submission of blood and archived tumor tissue sample from definitive surgery for next generation sequencing of the tumor. Tumor block is preferred however 14 slides + 1H&E can be submitted if necessary. NOTE: Due to possible false positives, ctDNA should not be drawn before completing radiation or less than 14 days from surgery if radiation is not required.
* Adequate laboratory values must be obtained within 28 days prior to study registration.

  * Hemoglobin (Hgb) ≥ 9.0 g/dL
  * Platelets ≥ 100 K/mm3
  * Absolute neutrophil count (ANC) ≥ 1.5 K/mm3
  * Calculated creatinine clearance of ≥ 50 cc/min using the Cockcroft-Gault formula
  * Bilirubin ≤ 1.5 ULN (except in participants with documented Gilbert's disease, who must have a total bilirubin ≤ 3.0 mg/dL)
  * Aspartate aminotransferase (AST, SGOT) ≤ 2.5 ULN
  * Alanine aminotransferase (ALT, SGPT) ≤ 2.5 ULN
* Women of childbearing potential and their partners and male subjects and their partners must be willing to use effective contraception (as outlined in protocol) from the time consent is signed until after protocol therapy discontinuation based on package insert or investigator brochure guidelines (See protocol for timeframes).
* Women of childbearing potential must have a negative urine or serum pregnancy test at screening and within 7 days prior to study registration. Women should be counseled regarding acceptable birth control methods to utilize. If prior to treatment after discussion with the subject it is felt by the treating physician there is a possibility the subject is pregnant a pregnancy test should be repeated. NOTE: Women are considered not of childbearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy), or they are postmenopausal for at least 12 consecutive months.
* Women must not be breastfeeding from the time of treatment initiation until the number of days after protocol therapy discontinuation based on package insert or investigator brochure guidelines (See protocol for timeframes).

Inclusion Criteria for Patients Assigned to Arm 1c ONLY

-Adequate laboratory values must be obtained within 21 days prior to starting arm therapy.

* Fasting total glucose ≤ 126 mg/dL
* HbA1C ≤ 5.7%
* Cholesterol < 300 mg/dL; 10.34 mmol/L
* Triglycerides < 300 mg/dL; 3.42 mmol/L

General Exclusion Criteria

* Clinically significant infections as judged by the treating physician.
* Stage IV (metastatic) disease, however no specific staging studies are required in the absence of symptoms or physical exam findings that would suggest distant disease.
* HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of registration are eligible for this trial. NOTE: Patients without a known history of being HIV positive do not require testing at screening. Patients who are known to be HIV positive will require testing as described to be eligible for this trial. Testing should be considered standard of care.
* Patients with evidence of chronic hepatitis B virus (HBV) infection, with undetectable HBV viral load within 6 months of registration are eligible for this trial. They should be on suppressive therapy, if indicated. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, the HCV viral load must be undetectable within 6 months of registration to be eligible for this trial. NOTE: Patients without a known history of being hepatitis positive do not require testing at screening. Patients who are known to be hepatitis positive will require testing as described to be eligible for this trial. Testing should be considered standard of care.
* Participants with unstable angina or a myocardial infarction within 12 months of study registration.
* Active second malignancy (except non-melanomatous skin cancer or incidental prostate cancer found on cystectomy): Active second malignancy is defined as a current need for cancer therapy or a high possibility (> 30%) of recurrence during the study. Previous contralateral breast cancer is allowable unless it meets "active" criteria as stated above.
* Inability to swallow pills.
* Evidence of significant uncontrolled concomitant disease that could affect compliance with the protocol, safety of participation, or interpretation of results. This includes significant liver disease (such as cirrhosis, uncontrolled major seizure disorder, or superior vena cava syndrome) or any other serious medical condition or abnormality in clinical laboratory tests that meet these criteria in the investigator's opinion.
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to any of the study medications being used in this study.
* Treatment with any investigational agent within 30 days prior to study registration.

Exclusion Criteria for Patients Assigned to Arm 1c ONLY

* Any concurrent ocular or intraocular condition (e.g., cataract or diabetic retinopathy) that, in the opinion of the investigator, would require medical or surgical intervention during the study period to prevent or treat vision loss that might result from that condition.
* Type 2 diabetes requiring ongoing systemic treatment at the time of study entry; or any history of Type 1 diabetes.
* Active inflammatory (e.g., uveitis or vitritis) or infectious (e.g., conjunctivitis, keratitis, scleritis, or endophthalmitis) conditions in either eye or history of idiopathic or autoimmune-associated uveitis in either eye.
* Symptomatic active lung disease, including pneumonitis
* History of or active inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis). Patients currently receiving immunosuppressants for inflammatory bowel disease (e.g., sulfasalazine) are considered to have active disease and are therefore ineligible.
* Any active bowel inflammation (including diverticulitis)
* Symptomatic hypercalcemia requiring continued use of bisphosphonate or denosumab therapy. Bisphosphonate and denosumab therapy for bone metastases or osteopenia/osteoporosis is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-08-24 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bryan P Schneider, MD, Principal Investigator — Indiana University
Locations (13):
- United States (13):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Georgetown University, Washington D.C., District of Columbia
  - Memorial Healthcare System, Hollywood, Florida
  - Miami Cancer Institute at Baptist Health, Inc., Miami, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Summit Health, Berkeley Heights, New Jersey
  - Novant Health Cancer Institute, Winston-Salem, North Carolina
  - Mays Cancer Center at UT Health San Antonio, San Antonio, Texas
  - University of Wisconsin, Madison, Wisconsin
  - Froedtert and The Medical College of Wisconsin, Milwaukee, Wisconsin
  - Advocate Aurora Research Institute (Illinois), Wauwatosa, Wisconsin
  - Aurora Health Care, Wauwatosa, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1c: ctDNA Positive Genomically Directed - PI3K Pathway: Arm 1c: Patients who are ctDNA-positive and harbor a genomic target. PI3K Pathway = inavolisib + capecitabine ---> +/- standard of care pembrolizumab
- Arm 2: ctDNA Positive -Standard of Care: Arm 2 subjects have plasma ctDNA positive but do not have a genomically driven treatment option. Treatment of physician's choice will be given with consideration for capecitabine and pembrolizumab. Dose, schedule and duration of treatment to be determined by treating physician.
  Capecitabine: Capecitabine 1000 mg/m2 BID Orally 14 days on and 7 days off Cycle = 21 days; Total of 8 cycles
  Pembrolizumab: Per standard of care.
- Arm 3: ctDNA Negative - Physician's Choice: Arm 3 subjects have plasma ctDNA negative. Treatment of patient and physician's choice will be given with consideration for capecitabine and pembrolizumab. Dose, schedule and duration of treatment to be determined by treating physician.
  Capecitabine: Capecitabine 1000 mg/m2 BID Orally 14 days on and 7 days off Cycle = 21 days; Total of 8 cycles
  Pembrolizumab: Per standard of care.
Period: Overall Study
Arm/Group | Arm 1c: ctDNA Positive Genomically Directed - PI3K Pathway | Arm 2: ctDNA Positive -Standard of Care | Arm 3: ctDNA Negative - Physician's Choice
Started | 1 | 5 | 46
Completed | 1 | 4 | 46
Not Completed | 0 | 1 | 0
Not completed — Eligibility criteria not meet | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 2: ctDNA Positive - Standard of Care: Arm 2 subjects have plasma ctDNA positive but do not have a genomically driven treatment option. Treatment of physician's choice will be given with consideration for capecitabine and pembrolizumab. Dose, schedule and duration of treatment to be determined by treating physician.
  Capecitabine: Capecitabine 1000 mg/m2 BID Orally 14 days on and 7 days off Cycle = 21 days; Total of 8 cycles
  Pembrolizumab: Per standard of care.
- Total: Total of all reporting groups
Arm/Group | Arm 1c: ctDNA Positive Genomically Directed - PI3K Pathway | Arm 2: ctDNA Positive - Standard of Care | Arm 3: ctDNA Negative - Physician's Choice | Total
Number analyzed (Participants) | 1 | 4 | 46 | 51
Age, Continuous [Median (Full Range); unit: years] | 47 [47 to 47] | 55 [30 to 61] | 51 [29 to 77] | 51 [29 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 46 | 51
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 5 | 5
  Not Hispanic or Latino | 1 | 4 | 41 | 46
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 12 | 13
  White | 1 | 3 | 33 | 37
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 4 | 46 | 51
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) from 0-5 that describes a patient's level of functioning where 0=Fully active, able to carry on all pre-disease performance without restriction and 5=Dead:
  1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work, 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours.
  Participants
    ECOG = 0 | 1 | 2 | 37 | 40
    ECOG = 1 | 0 | 2 | 8 | 10
    Missing | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: ARM 1c: Disease Free Survival (DFS) at 2 Years
Description: DFS is defined as the duration of time from arm assignment to time of a DFS event, defined as local failure (invasive), regional failure, distant failure, contralateral breast cancer (invasive or non-invasive), or death from any cause.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1c: ctDNA Positive Genomically Directed - PI3K Pathway
Number analyzed (Participants) | 1
Percentage of participants | 100 [100 to 100]

2. Secondary Outcome: ARM 2: Disease Free Survival (DFS) at 2 Years
Description: as for outcome 1
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 2: ctDNA Positive - Standard of Care
Number analyzed (Participants) | 4
Percentage of participants | 0 [NA to NA] — Not enough events occur to calculate 95% confidence interval.

3. Secondary Outcome: ARM 3:Disease Free Survival (DFS) at 2 Years
Description: as for outcome 1
Time Frame: 2 years
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoint Disease free survival was defined as all patients who received at least one dose of study treatment and have had at least one post baseline disease assessment or die before first assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 3: ctDNA Negative - Physician's Choice
Number analyzed (Participants) | 40
Percentage of participants | 40.2 [11.7 to 67.9]

4. Secondary Outcome: Overall Disease Free Survival (DFS)
Description: Comparison of overall DFS in Arms 1c, 2, 3. DFS is defined as the duration of time from arm assignment to time of a DFS event such as local failure (invasive), regional failure, distant failure, contralateral breast cancer (invasive or non-invasive), or death from any cause
Time Frame: Up to 29 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1c: ctDNA Positive Genomically Directed - PI3K Pathway | Arm 2: ctDNA Positive - Standard of Care | Arm 3: ctDNA Negative - Physician's Choice
Number analyzed (Participants) | 1 | 4 | 40
Months | 27.7 [NA to NA] — Not enough events occur to calculate 95% confidence interval | 8.1 [2.9 to NA] — Not enough events occur to calculate upper 95% confidence interval | 23.1 [16.7 to NA] — Not enough events occur to calculate upper 95% confidence interval

5. Secondary Outcome: Overall Distant Disease Free Survival (DDFS)
Description: DDFS is defined as the duration of time from arm assignment to time of recurrence of breast cancer outside the breast and/or death from any cause.
Time Frame: Up to 29 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1c: ctDNA Positive Genomically Directed - PI3K Pathway | Arm 2: ctDNA Positive - Standard of Care | Arm 3: ctDNA Negative - Physician's Choice
Number analyzed (Participants) | 1 | 4 | 40
Months | 27.7 [NA to NA] — Not enough events occur to calculate 95% confidence interval | 8.1 [3.1 to NA] — Not enough events occur to calculate upper 95% confidence interval | 23.1 [18.8 to NA] — Not enough events occur to calculate upper 95% confidence interval

6. Secondary Outcome: 1-year Disease Free Survival (DFS)
Description: Compare 1-year DFS in Arms 1c, 2, 3. DFS is defined as the duration of time from arm assignment to time of a DFS event, defined as local failure (invasive), regional failure, distant failure, contralateral breast cancer (invasive or non-invasive), or death from any cause
Time Frame: 1 year
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1c: ctDNA Positive Genomically Directed - PI3K Pathway | Arm 2: ctDNA Positive - Standard of Care | Arm 3: ctDNA Negative - Physician's Choice
Number analyzed (Participants) | 1 | 4 | 40
Percentage of participants | 100 [100 to 100] | 0 [NA to NA] — Not enough events occur to calculate 95% confidence interval. | 79.8 [59.9 to 90.6]

7. Secondary Outcome: Overall Survival (OS) at 5 Year
Description: Overall survival is defined as the time from date of treatment start until death from any cause.
Time Frame: 5 years
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoint 5 -years Overall survival was defined as all patients who received at least one dose of study treatment and have follow-up up to 5 years. Because of the early termination, 5-year overall survival was not reached by any subjects.
Arm/Group | Arm 1c: ctDNA Positive Genomically Directed - PI3K Pathway | Arm 2: ctDNA Positive - Standard of Care | Arm 3: ctDNA Negative - Physician's Choice
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events (regardless of relationship with study drug) will be assessed using the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) criteria v5
Time Frame: Up to 16 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1c: ctDNA Positive Genomically Directed - PI3K Pathway | Arm 2: ctDNA Positive - Standard of Care | Arm 3: ctDNA Negative - Physician's Choice
Number analyzed (Participants) | 1 | 4 | 46
Participants | 1 | 3 | 42

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored up to a maximum of 35 months. Serious Adverse Events and Other (Not Including Serious) Adverse Events were monitored from time of initiation of study drug until 30 days after discontinuation of study drug(s) or until a new anti-cancer treatment starts, up to a maximum of 16 months.
Arm/Group | Arm 1c: ctDNA Positive Genomically Directed - PI3K Pathway | Arm 2: ctDNA Positive - Standard of Care | Arm 3: ctDNA Negative - Physician's Choice
All-Cause Mortality (participants affected / at risk) | 0/1 | 1/4 | 4/46
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/4 | 3/46
Other Adverse Events (participants affected / at risk) | 1/1 | 3/4 | 33/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1c: ctDNA Positive Genomically Directed - PI3K Pathway (N=1) | Arm 2: ctDNA Positive - Standard of Care (N=4) | Arm 3: ctDNA Negative - Physician's Choice (N=46)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
NERVOUS SYSTEM DISORDERS - OTHER, SPECIFY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1c: ctDNA Positive Genomically Directed - PI3K Pathway (N=1) | Arm 2: ctDNA Positive - Standard of Care (N=4) | Arm 3: ctDNA Negative - Physician's Choice (N=46)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2)
ANEMIA (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (1)
ANOREXIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2)
ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
BREAST PAIN (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
CHEST WALL NECROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
DIARRHEA (Gastrointestinal disorders) | 1 (3) | 0 (0) | 8 (11)
DRY EYE (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
EDEMA LIMBS (General disorders) | 1 (1) | 0 (0) | 0 (0)
EYELID FUNCTION DISORDER (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 1 (6) | 0 (0) | 5 (7)
FEVER (General disorders) | 1 (1) | 0 (0) | 0 (0)
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1 (3) | 1 (1) | 0 (0)
HYPOKALEMIA (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (1)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
INSOMNIA (Psychiatric disorders) | 1 (4) | 0 (0) | 0 (0)
JOINT RANGE OF MOTION DECREASED (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
LYMPH NODE PAIN (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
LYMPHEDEMA (Vascular disorders) | 1 (3) | 0 (0) | 0 (0)
MUCOSITIS ORAL (Gastrointestinal disorders) | 1 (6) | 0 (0) | 5 (5)
NAUSEA (Gastrointestinal disorders) | 1 (5) | 0 (0) | 6 (6)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) - OTHER, SPECIFY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
PAIN (General disorders) | 1 (2) | 0 (0) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
PALMAR-PLANTAR ERYTHRODYSESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 1 (9) | 0 (0) | 12 (16)
PALPITATIONS (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 (4) | 0 (0) | 3 (3)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
SEIZURE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 (1) | 0 (0) | 2 (2)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (3) | 0 (0) | 1 (1)
WOUND INFECTION (Infections and infestations) | 1 (5) | 0 (0) | 0 (0)
CD4 LYMPHOCYTES DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
LYMPHOCYTE COUNT DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
WEIGHT GAIN (Investigations) | 0 (0) | 1 (1) | 1 (1)
WHITE BLOOD CELL DECREASED (Investigations) | 0 (0) | 1 (1) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
BLURRED VISION (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
CHEST WALL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
COLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
DYSURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
EDEMA CEREBRAL (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
EYE DISORDERS - OTHER, SPECIFY (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
HEPATOBILIARY DISORDERS - OTHER, SPECIFY (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
HOT FLASHES (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
INVESTIGATIONS - OTHER, SPECIFY (Investigations) | 0 (0) | 0 (0) | 1 (1)
METABOLISM AND NUTRITION DISORDERS - OTHER, SPECIFY (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER - OTHER, SPECIFY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OBESITY (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
VAGINAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
WEIGHT LOSS (Investigations) | 0 (0) | 0 (0) | 2 (2)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-14): https://cdn.clinicaltrials.gov/large-docs/64/NCT04849364/Prot_SAP_000.pdf